CLINICAL TRIAL: NCT01659853
Title: A Multicenter, Randomized, Controlled, Double-masked, Crossover Design Study to Compare Efficacy and Assess Safety of CD07805/47 Gel 0.5% Applied Once Daily vs Azelaic Acid Gel 15% Applied Twice Daily in Subjects With Erythema of Rosacea
Brief Title: Efficacy and Safety Study Comparing CD07805/47 Gel 0.5% to Azelaic Acid Gel 15% in Subjects With Erythema of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US10219
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2014-03

CONDITIONS: Erythema; Rosacea
MeSH Terms: conditions — Erythema; Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Study (Experimental): In this crossover study of CD07805/47 gel 0.5%/CD07805/47 Vehicle and azelaic acid gel 15%, 70 subjects were randomly assigned to treatment sequence.
  During Period 1 (15 days), 35 subjects received topical CD07805/47 gel 0.5% in the morning and topical CD07805/47 gel vehicle in the evening, and 35 received topical azelaic acid gel twice daily according to FDA approved prescribing information. Subjects crossed over to the other treatment in Period 2 (15 days).
  Interventions: Drug: CD07805/47 gel 0.5%/CD07805/47 Vehicle; Drug: azelaic acid gel 15%

INTERVENTIONS:
Drug: CD07805/47 gel 0.5%/CD07805/47 Vehicle — To maintain masking, CD07805/47 gel 0.5% will be administered along with CD07805/47 gel vehicle.
  During each treatment period (baseline to Day 15):
  CD07805/47 gel 0.5%, topical, once daily and CD07805/47 gel vehicle, topical, once daily
  Other Names: brimonidine tartrate gel 0.5%; brimonidine tartrate gel vehicle
Drug: azelaic acid gel 15% — During each treatment period (baseline to Day 15): azelaic acid gel 15%, topical, twice daily
  Other Names: Finacea® gel 15%

SUMMARY:
The purpose of this study is to compare the efficacy and assess the safety of CD07805/47 gel 0.5% applied topically once daily versus azelaic acid gel 15% applied topically twice daily in subjects with moderate to severe facial erythema of rosacea.

DETAILED DESCRIPTION:
Adult subjects with moderate to severe facial erythema of rosacea who meet inclusion/exclusion criteria will be randomized at Baseline/Visit 1 in a 1:1 ratio to receive either CD07805/47 gel 0.5% once daily or azelaic acid gel 15% twice daily for 15 days. Following an appropriate washout period, subjects will then switch treatments and use the second investigational product as instructed for 15 days (according to the subject's randomization scheme). Subjects will re-qualify based upon inclusion/exclusion prior to Period 2 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female aged 18 years or older.
2. Subject has a clinical diagnosis of facial rosacea.
3. Subject has a clinician's assessment score of moderate to severe erythema prior to enrollment.
4. Subject has a self assessment score of moderate to severe redness prior to enrollment.
5. Subjects with none to mild facial inflammatory lesions of rosacea prior to enrollment.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing or planning a pregnancy during the study.
2. Subjects with a condition or who are in a situation, which in the Investigator's opinion may put a subject at risk, may confound study results, or may interfere with a subject's participation in the study.
3. Subjects with conditions causing facial erythema which would confound the assessment of treatment.
4. Subjects who are taking or have recently taken medications known to have interactions with α2-adrenergic agonists.
5. Subjects with known allergies or sensitivities to one of the components of the investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Gottschalk, MD, Study Director — Galderma R&D
Locations (4):
- United States (4):
  - Hudson Dermatology, Evansville, Indiana
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - DermResearch, Inc, Austin, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- CD07805/47 Gel 0.5% and Vehicle, Then Azelaic Acid Gel 15%; Azelaic Acid Gel 15%, Then CD07805/47 Gel 0.5% and Vehicle: Subjects were randomly assigned to treatment sequence.
  Subjects who received CD07805/47 gel 0.5% and CD07805/47 gel vehicle during Period 1 (baseline to Day 15) will switch to azelaic acid gel in Period 2.
  Subjects who received azelaic acid gel 15% during Period 1 (baseline to Day 15) switched to CD07805/47 gel 0.5% and CD07805/47 gel vehicle in period 2.
  Subjects assigned to brimonidine tartrate gel 0.5% applied it once daily in the morning and applied brimonidine tartrate gel vehicle once daily in the evening. Subjects assigned to azelaic acid gel 15% applied it twice daily according to FDA approved prescribing information.
Period: Treatment Period 1
Arm/Group | CD07805/47 Gel 0.5% and Vehicle, Then Azelaic Acid Gel 15% | Azelaic Acid Gel 15%, Then CD07805/47 Gel 0.5% and Vehicle
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Washout , 3 to 7 Days
Arm/Group | CD07805/47 Gel 0.5% and Vehicle, Then Azelaic Acid Gel 15% | Azelaic Acid Gel 15%, Then CD07805/47 Gel 0.5% and Vehicle
Started | 35 | 35
Completed | 33 | 35
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Treatment Period 2
Arm/Group | CD07805/47 Gel 0.5% and Vehicle, Then Azelaic Acid Gel 15% | Azelaic Acid Gel 15%, Then CD07805/47 Gel 0.5% and Vehicle
Started | 33 | 35
Completed | 33 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants were randomly assigned to treatment sequence.
  Subjects who received CD07805/47 gel 0.5% and CD07805/47 gel vehicle during Period 1 (baseline to Day 15) switched to azelaic acid gel in Period 2.
  Subjects who received azelaic acid gel 15% during Period 1 (baseline to Day 15) switched to CD07805/47 gel 0.5% and CD07805/47 gel vehicle in Period 2.
  Subjects assigned to brimonidine tartrate gel 0.5% applied it once daily in the morning and applied brimonidine tartrate gel vehicle once daily in the evening. Subjects assigned to azelaic acid gel 15% applied it twice daily according to FDA approved prescribing information.
Arm/Group | Overall Study
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 70
Fitzpatrick skin type [Number; unit: participants] — Fitzpatrick Skin Type Classification Scale I, always burns easily; never tans II, always burns easily; tans minimally and with difficulty III, burns minimally; tans gradually and uniformly (light brown) IV, burns minimally; always tans well (moderate brown) V, rarely burns; tans very easily (dark brown) VI, never burns, tans very easily (black)
  participants
    I | 6
    II | 35
    III | 24
    IV | 4
    V | 1
    VI | 0
Skin type [Number; unit: participants]
  Dry | 14
  Normal | 33
  Oily | 6
  Combination | 17

OUTCOME MEASURES:

1. Primary Outcome: Composite Success
Description: Composite Success, defined as a 2-grade improvement at 6 hours on both the clinician's and subject's erythema assessments at the end of each treatment period
Time Frame: Hour 6 on Day 15
Population: A carryover effect was observed from Period 1 to Period 2. Therefore, as specified in the protocol, only the Period 1 results were analyzed.
Measure: Number; unit: percentage of subjects
Groups:
- CD07805/47 Gel 0.5% and Vehicle; Azelaic Acid Gel 15%: Participants were randomly assigned to treatment sequence. Thirty-five subjects received CD07805/47 gel 0.5% and 35 received azelaic acid gel in Period 1.
  A carryover effect was observed from Period 1 to Period 2. Therefore, as specified in the protocol, only the Period 1 results were analyzed.
Arm/Group | CD07805/47 Gel 0.5% and Vehicle | Azelaic Acid Gel 15%
Number analyzed (Participants) | 35 | 35
percentage of subjects | 14.3 | 5.7

2. Secondary Outcome: Onset of Action
Description: Onset of action, defined as an improvement on both the clinician's and subject's erythema assessments at 30 minutes post baseline application
Time Frame: 30 minutes after baseline treatment application on Day 15
Population: A carryover effect was observed from Period 1 to Period 2. Therefore, as specified in the protocol, only the Period 1 results were analyzed. All 70 enrolled subjects were analyzed for efficacy.
Measure: Number; unit: percentage of subjects
Groups:
- CD07805/47 Gel 0.5 and Vehicle; Azelaic Acid 15%: Participants were randomly assigned to treatment sequence. Thirty-five subjects received CD07805/47 gel 0.5% and 35 received azelaic acid gel in Period 1.
  A carryover effect was observed from Period 1 to Period 2. Therefore, as specified in the protocol, only the Period 1 results were analyzed.
Arm/Group | CD07805/47 Gel 0.5 and Vehicle | Azelaic Acid 15%
Number analyzed (Participants) | 35 | 35
percentage of subjects | 31.4 | 29.4

ADVERSE EVENTS:
Time Frame: 15 days
Description: Two subjects in the CD07805/47 group in period 1 did not enter period 2 (1 AE and 1 protocol violation). Therefore, 70 subjects received CD07805/47 and 68 received azelaic acid.
Groups:
- CD07805/47 Gel 0.5 and Vehicle; Azelaic Acid 15%: Participants were randomly assigned to treatment sequence.
  Subjects who received CD07805/47 gel 0.5% and CD07805/47 gel vehicle during Period 1 (baseline to Day 15) switched to azelaic acid gel in Period 2.
  Subjects who received azelaic acid gel 15% during Period 1 (baseline to Day 15) switched to CD07805/47 gel 0.5% and CD07805/47 gel vehicle in Period 2.
  Subjects assigned to brimonidine tartrate gel 0.5% applied it once daily in the morning and applied brimonidine tartrate gel vehicle once daily in the evening. Subjects assigned to azelaic acid gel 15% applied it twice daily according to FDA approved prescribing information.
Arm/Group | CD07805/47 Gel 0.5 and Vehicle | Azelaic Acid 15%
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 19/70 | 27/68
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD07805/47 Gel 0.5 and Vehicle (N=70) | Azelaic Acid 15% (N=68)
Medication residue (General disorders) | 0 (0) | 9 (9)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 15 (20) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (11)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
A significant period effect was observed for CEA indicating there was carryover from period 1 to period 2. Therefore, as stated a priori in the protocol, only data from period 1 were used to analyze efficacy. All safety data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days